CLINICAL TRIAL: NCT02283398
Title: The CARE-TAVI Study: Cardioprotective Effect of Remote Ischemic Preconditioning in Patients Undergoing Transcatheter Aortic Valve Implantation
Brief Title: Cardioprotective Effect of RIPC in Patients Undergoing TAVI
Acronym: CARE-TAVI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: administrative issues
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CARE-TAVI
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Effectivity of RIPC in Outcomes of TAVI Procedure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- with RIPC (Experimental): RIPC will be induced with three cycles of inflation of a blood-pressure cuff on the left arm to 200 mm Hg for 5 min, followed by 5 min of reperfusion while cuff deflated
  Interventions: Procedure: RIPC
- without RIPC (Sham Comparator): the cuff will be placed around the left arm without being inflated
  Interventions: Other: without RIPC

INTERVENTIONS:
Other: without RIPC — the cuff will be placed around the left arm without being inflated
  Other Names: no remote ischemic preconditioning
  Arms: without RIPC
Procedure: RIPC — RIPC will be induced with three cycles of inflation of a blood-pressure cuff on the left arm to 200 mm Hg for 5 min, followed by 5 min of reperfusion while cuff deflated
  Other Names: remote ischemic preconditioning
  Arms: with RIPC

SUMMARY:
We aim to investigate whether RIPC (remote ischemic preconditioning) is effective in the TAVI setting to reduce post-procedural myocardial damage and improve patient outcome. Accordingly, we aim to investigate whether RIPC can be introduced as an integral part of the TAVI procedure, in order to reduce post-procedural myocardial damage and potentially improve patient outcome.

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) is associated to myocardial injury, defined as post-procedural cardiac troponin (cTn) elevation. Earlier experiences have shown that myocardial damage can be encountered in a percentage of patients that varies from 1.5% to 17%, depending on the access route (transfemoral and transapical, respectively). The degree of rise in cTn after TAVI emerged as an independent predictor of mortality.

Remote ischaemic preconditioning (RIPC) consists of brief episodes of ischaemia applied to remote organs or tissues and has shown to result in a significant reduction in postoperative troponin levels in cardiac and non-cardiac surgery patients. Lately, growing evidence suggests that post-procedural troponin decreases due to RIPC application protocols protocols and is associated with improved outcome.

The patients will be divided into two Groups. In Group 1, RIPS will be induced with three cycles of Inflation of a blood-pressure cuff on the left arm to 200 mmHg for 5 min., followed by 5 min. of reperfusion while the cuff is deflated. In controls (Group 2), the cuff will be placed around the left arm without being inflated.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective TAVI following Heart Team discussion
* Stable hemodynamic conditions without circulatory support or catecholamines

Exclusion Criteria:

* Myocardial infarction at least 3 months before enrollment
* Stroke/TIA at least 3 months before enrollment
* Severe chronic kidney disease (defined as a baseline serum creatinine of > 1.5 mg/dl or an estimated glomerular filtration rate (eGFR) of 60 ml/min/1.73 m2 )
* PCI at least 3 months before enrollment
* Abnormal (>99th percentile of laboratory cut-off) baseline values of biomarkers of myocardial ischemia (i.e. TnT, CK-MB)
* Abnormal NSE values at baseline (local laboratory cut-off values)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
post-procedural myocardial injury, defined by the geometric mean (95% CI) of the area under the curve (AUC) for cTnT | 72 hours after intervention
  Change in cardiac troponine T (cTnT)

SECONDARY OUTCOMES:
Post-procedural myocardial injury | 72 hours after intervention
  defined by the geometric mean (95% CI) of the area under the curve (AUC) for CK-MB
Post-procedural acute kidney injury | 72 hours after intervention
  defined according to the VARC 2 criteria
Post-procedural brain injury | 72 hours after intervention
  defined by the geometric mean (95% CI) of the area under the curve (AUC) for NSE
composite of major adverse cardiac and cerebrovascular events | discharge, at 30 days and at 1 year
  including death, postoperative myocardial infarction and cerebrovascular accident or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Naber, PD Dr. med., Principal Investigator — Elisabeth-Krankenhaus Essen, Klinik für Kardiologie und Angiologie
Locations (3):
- Germany (3):
  - Klinikum Dortmund, Medizinische Klinik Mitte - Kardiologie, Dortmund
  - Evangelisches Klinikum Niederrhein, Kardiologie, Duisburg
  - Klinikum Karlsruhe, Karlsruhe